CLINICAL TRIAL: NCT00213668
Title: Effect of Glutamine on Gastric Emptying and Length of Parenteral Nutrition in Premature Neonates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2000/111/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Enteral Feeding
Keywords: glutamine; premature neonate; gastric emptying
MeSH Terms: conditions — Premature Birth | interventions — Glutamine; alanylglutamine

INTERVENTIONS:
Dietary Supplement: glutamine (dipeptiven)

SUMMARY:
This study investigates the effects of enterally supplied glutamine on gastric emptying, intestinal transit, age of total enteral nutrition and age at the end of hospitalisation. Forty neonates, aged at least 2 days and free of acute illness participate in a prospective, randomised, double-blind study. All are fed with parenteral and enteral nutrition enriched with glutamine (0.7 g/kg/per day, group 1) or isonitrogenous control (group 2). Gastric emptying is analysed by sequential measure of intragastric residue by diluted polyethylene glycol (PEG) 4000. Intestinal transit is analysed by Rouge Carmin test.

ELIGIBILITY:
Inclusion Criteria:

* Premature neonates aged 30-33 weeks of gestational age
* Aged at least 2 days and no more than 10 days
* Free of acute illness
* Written informed consent is obtained from the parent prior to enrolment.

Exclusion Criteria:

* Premature infants with respiratory (fraction of inspired oxygen [FiO2] > 30%), or cardiovascular, liver, intestinal or acute diseases
* Premature infants with congenital syndrome

Ages: 2 Days to 10 Days | Sex: All
Age Groups: Child
Dates: Start 2002-04

PRIMARY OUTCOMES:
gastric emptying | at day 0, day 1, day 7 and day 14 of enteral nutrition enriched by glutamine or isonitrogenous product

SECONDARY OUTCOMES:
intestinal transit | at day 1 and day 14 of enteral nutrition enriched by glutamine or isonitrogenous product
date and duration of arrest of nutrition if necessary
age of total enteral nutrition
age at the end of hospitalization
variation of cholescystokinin and gastrin postprandial concentration | at day 0 and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mercier, MD, Principal Investigator — CHU Rouen
Locations (1):
- CHU-Rouen, Rouen, France